CLINICAL TRIAL: NCT06376123
Title: Nomogram for Prediction of Alveolo-arterial Gradient During One-lung Ventilation
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nıgar Kangarlı, Medical Doctor, Anesthesiologist, Bezmialem Vakif University
Other Study IDs: Nkangarli001
Record Dates: First submitted 2024-04-17; First posted 2024-04-19 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: One-lung Ventilation
Keywords: One lung ventilation; Alveolo-arterial gradient; Nomograms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Video assisted thoracoscopic surgery patients: Patients, assigned for elective lung surgery, older than 18 years and requiring one-lung ventilation.

SUMMARY:
The cause of hypoxia during one-lung ventilation is a common anaesthetic problem seen during thoracic surgery and is associated with increased fraction of shunted blood. This shunt occurs because the lung not participating in respiration stops saturating the blood with oxygen. The importance of our study is to collect some of the patient's parameters on a nomogram in the preoperative period, to predict the shunt fraction that will occur during one-lung ventilation and to make preparations and interventions accordingly.

DETAILED DESCRIPTION:
The shunt that occurs during one lung ventilation varies for each patient and depends on many parameters. In this study, our aim was to predict the level of shunting during anaesthesia using readily available preoperative data. It is important to predict the hypoxia that will develop due to the shunt and to plan the methods that can be applied to reduce the shunt in terms of patient safety. One of the most reliable data reflecting the shunt level is the gradient of alvelo- arterial oxygen concentration. The calculation of alveolo-arterial oxygen gradient (A-a O2 gradient) is based on easily accessible parameters (pO2, pCO2, FiO2, age). The secondary aim of the study is to follow how the A-a O2 gradient (oxygen difference between alveolar and arterial blood) changes over time during surgery.

Demographic data, planned operation, comorbidities, side of surgery, ASA score, preoperative haemoglobin level, FEV1 (forced expiratory volume in 1 minute), FEV1/FVC (forced expiratory volume in 1 minute/forced vital capacity) ratio and EF (ejection fraction) will be recorded before surgery.FEV1, FEV1/FVC ratio values will be measured by spirometry test. Spirometry is a preoperative test routinely performed in all patients undergoing one lung ventilation. EF will be measured by preoperative echocadiography, which is also performed during the preoperative preparation of all patients scheduled for lung surgery. Patients undergoing VATS (video-assisted thoracoscopy) surgery with planned lung resection, lobectomy, pulmonectomy, segmentectomy etc. will be included in the study and all will be operated in the lateral decubitus position.

Once the patient is on the operating table, routine haemodynamic monitoring (heart rate, non-invasive blood pressure and blood oxygen saturation) will be performed.

The patient will then have an arterial cannula inserted for invasive arterial monitoring. It is a routine practice in major surgeries for blood gas monitoring, haemorrhage monitoring and monitoring of sudden blood pressure fluctuations. After insertion of the arterial cannula, blood gas will be taken in room air and arterial pO2 (partial oxygen pressure), arterial pCO2 (partial carbon dioxide pressure) and arterial SpO2 (oxygen saturation) will be recorded. At the same time, a venous blood sample (from any vein in the upper limb) will be taken in room air and vSpO2 (venous blood oxygen saturation) will be recorded. The difference between SpO2 of arterial and venous blood is determined as Delta-SpO2 and is a specific parameter of this study.

All patients will undergo general anaesthesia and orotracheal intubation with a double lumen tube.

For anaesthesia induction, 1 mcg/kg fentanyl, 2 mg/kg propofol and 0.6 mg/kg rocuronium will be administered .After adequate mask ventilation and complete muscle relaxation, a double lumen intubation tube will be placed into the trachea by direct laryngoscopy. After the position of the tube and whether it is in the correct bronchus is supported by bronchoscopy, the patient will be connected to the mechanical ventilator and lateral decubitus (provided that the side to be operated on remains on top) will be given. Ventilator parameters will be selected the same for all patients. During two-lung ventilation, tidal volume 8 ml/kg, respiratory rate 12, peep 5, and FiO2 (fraction of inspired oxygen) = 60%. During one-lung ventilation, tidal volume will be set to 6 ml/min, respiratory rate 15, peep 5, and FiO2 = 70%. All patients will be ventilated in volume control mode.

At this stage, EtCO2 (end-tidal carbon dioxide) will be measured separately in both lungs. For this, first the airway from the lower lung will be clamped and the EtCO2 value will be recorded (dEtCO2 - dependent lung EtCO2). Then, vice versa, the airway from the lower lung will be clamped and the EtCO2 value obtained (ndEtCO2 - non-dependent lung EtCO2) will be recorded. The difference between these two values, D-EtCO2 (delta - end-tidal carbon dioxide) will be added to the data.

After these steps, one-lung ventilation will be started and the first A-a oxygen gradient will be recorded 30 minutes after initiation of OLV. The consequent calculations of OLV will be made every 30 minutes until the end of the surgery. The consequent measurements are necessary for estimation the A-a gradient change over time.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective VATS surgery.
* Age over 18 years.
* ASA 1-4 patients.

Exclusion Criteria:

* Patient refusal.
* Age below 18 years.
* Conditions that may impair oxygen diffusion: pulmonary oedema, fibrosis, interstitial lung disease, pneumonia.
* Emergency surgery.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes patients with pulmonary diseases, indicated for surgery. Among them are pulmonectomy, segmentectomy, lobectomy or wedge resections. All these types of surgery require one-lung (non-operating lung) ventilation. The patients should be electively operated, aged more that 18 years and must have no other pulmonary conditions (like fibrosis, pneumonia, lung oedema or interstitial lung disease) that could interfere with Alveolo-arterial gradient calculations.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Alveolo-arterial gradient | 30 mins after intubation
  The gradient of oxygen concentration between alveoli and arterial blood, achieved after patient switch from double lung to one lung lung ventilation. Is calculated automatically, based on oxygen tension in arterial and venous blood, which measured by blood gas analysis.

SECONDARY OUTCOMES:
Alveolo-arterial gradient change | After switching to one lung ventilation
  The gradient of oxygen concentration between alveoli and arterial blood, achieved after patient switch from double lung to one lung lung ventilation. It is measured be blod gas analysis. The secondary outcome involves the changes of the first outcome throughout the surgery and is measured every 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Nigar Kangarli, MD, Principal Investigator — Anesthesiology and Reanimation Department, Specialist
Locations (1):
- Bezmialem Vakif University Dragos Hospital, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parab SY, Chatterjee A, Saxena RS. The utility of gradient of end-tidal carbon dioxide between two lungs in lateral decubitus position in predicting a drop in oxygenation during one-lung ventilation in elective thoracic surgery- A prospective observational study. Indian J Anaesth. 2021 Oct;65(10):744-749. doi: 10.4103/ija.ija_591_21. Epub 2021 Oct 29. PMID 34898701
- [Background] Karzai W, Schwarzkopf K. Hypoxemia during one-lung ventilation: prediction, prevention, and treatment. Anesthesiology. 2009 Jun;110(6):1402-11. doi: 10.1097/ALN.0b013e31819fb15d. PMID 19417615
- [Background] Alday E, Nieves JM, Planas A. Oxygen Reserve Index Predicts Hypoxemia During One-Lung Ventilation: An Observational Diagnostic Study. J Cardiothorac Vasc Anesth. 2020 Feb;34(2):417-422. doi: 10.1053/j.jvca.2019.06.035. Epub 2019 Jun 28. PMID 31362907